CLINICAL TRIAL: NCT02539524
Title: Effects of Yoga Respiratory Exercises on Clinical Impact, and Psychosocial Aspects in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Yoga on Clinical Impact and Psychosocial Aspects of COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Danilo Forghieri Santaella, Ph.D., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 102838/2014
Record Dates: First submitted 2015-08-28; First posted 2015-09-03 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Pulmonary Obstructive Disease
Keywords: clinical impact; anxiety; quality of life; Yoga
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary Rehabilitation Group (Active Comparator): Pulmonary Rehabilitation Group Intervention consisted of 12-week pulmonary rehabilitation. Two 1 hour sessions a week, consisting of: 30 min of aerobic training followed by resistance exercises for upper and lower limbs.
  Interventions: Other: Pulmonary Rehabilitation
- Yoga Group (Experimental): Yoga Bhastrika Pranayama breathing exercises consisted of: 12-week pulmonary rehabilitation (two 1 hour sessions a week, consisting of: 30 min of aerobic training followed by resistance exercises for upper and lower limbs). After each pulmonary rehabilitation session, participants of this group performed 10 bhastrika pranayama breathing exercises (1 bhastrika is formed by 20 kapalabhati followed by 1 surya bedhana - described earlier).
  Interventions: Other: Yoga bhastrika pranayama breathing exercise

INTERVENTIONS:
Other: Yoga bhastrika pranayama breathing exercise — Bhastrika Pranayama is formed by a set of 20 nasal forced and rapid expirations, followed by passive nasal inspirations, followed by 1 alternate nasal breath which always begins through the right nostril, and has a retention between intake and outflow. The set of this breathing exercise is supposed to bring respiratory relief.
  Arms: Yoga Group
Other: Pulmonary Rehabilitation — Pulmonary Rehabilitation Group Intervention consisted of 12-week pulmonary rehabilitation. Two 1 hour sessions a week, consisting of: 30 min of aerobic training followed by resistance exercises for upper and lower limbs.
  Arms: Pulmonary Rehabilitation Group

SUMMARY:
The aim of this study is to investigate weather the breathing exercises of Yoga are effective in altering clinical impact, anxiety, depression and quality of life in Chronic Obstructive Pulmonary Disease patients.

DETAILED DESCRIPTION:
Introduction According to the Global Initiative for Chronic Lung Disease (GOLD), chronic obstructive pulmonary disease (COPD) is a common, preventable and treatable disease, characterized by a persistent not totally reversible limitation of air flow, with a progressively characteristic associated to the increase of inflammatory lungs and air pathways reactions to gas and harmful particles. It is one of the main morbid-mortality causes world wide and, thus, a social health matter. Dyspnoea is a recurrent stressful symptom of COPD, and is usually followed by anxiety, depression, and decreased quality of life.

Some studies have addressed the tolerance of yoga breathing exercises by COPD patients, and some have indeed found a decreased functional load of dyspnoea in such patients.

Thus, the aim of this study is to investigate the effects of the regular practice (training) of respiratory Yoga exercises (pranayamas) on the clinical impact and psychosocial aspects: anxiety, depression and quality of life in COPD patients as a complementary therapy to pulmonary rehabilitation.

Methods Participants Diagnosed COPD patients will be recruited from the Pulmonary Rehabilitation Ambulatory of the Clinical Hospital of the Faculty of Medicine of the University of São Paulo (HC-FMUSP). All participants will give written consent to participate of the study, and will be able to exit the study at any point without having to explain the reason.

Sample Size Calculation Based on effect expected proportion in controls of 0.05, assuming an odds ratio of 25, in a confidence level of 0.95, and a power of 0.8, the sample size for each group was 9, in a total sample size (both groups) of 18 participants.

Experimental Design This is a randomized controlled prospective clinical trial, with two groups: pulmonary rehabilitation for control group (PRG) and pulmonary rehabilitation plus Yoga group (YG).Randomization was carried out by numbered paper draw: 20 papers numbered from 1-20 were put in a bag from which participants took 1 paper each. Even numbers indicated PRG and odd ones indicated YG. Medication will not altered during study. Both groups will perform a 12-week pulmonary rehabilitation program, besides that, YG will perform 24 Yoga breathing sessions (2 times a week). Participants of both groups will answer questionnaires to evaluate clinical impact, anxiety, depression and quality of life at study entry and after 12 weeks.

Yoga Breathing Exercises Breathing exercises will be based on traditional Hatha Yoga texts (Hathapradipika and Gheranda Samhita). The chosen exercise was bhastrika pranayama (kapalabhati followed by surya bedhana). Kapalabhhati consists basically of 20 fast and vigorous abdominal contractions for expiration, followed by immediate and maximal relaxation of these muscles for inspiration, and surya bedhana is a slow inspiration through the right nostril, followed by a comfortable apnoea for the same time of air intake, and a slower yet comfortable expiration through the left nostril. During training, participants will be considered at peak training when they are able to perform 10 sets of bhastrika.

Pulmonary Rehabilitation will consist of 30 minutes of aerobic training (cycloergometer or treadmill) followed by resistance exercises for lower and upper limbs.

Evaluations Clinical impact of COPD will be accessed by the COPD Assessment Test; anxiety will be evaluated by Hospital Anxiety and Depression Scale; Quality of Life will be accessed by the self-reported Chronic Respiratory Questionnaire.

Statistical Analysis Intra-group comparisons between moments (pre vs. post treatment) will be done using a paired Student T-test (repeated measures). While inter-groups comparisons (PRG vs. YG) will be done using the independent measures Student T-test. Significance will be accepted when p<0.05. SPSS v.21 software will be used to process analysis.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosed classified as B, C or D according to the Global Initiative for Obstructive Lung Disease (GOLD);
* Optimized medical treatment.

Exclusion Criteria:

* Any other lung disease;
* Home use of oxygen therapy;
* Respiratory Yoga exercise training in the last 2 years;
* Current smokers.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in COPD Clinical Impact | Baseline and 12 weeks
  Evaluated by COPD Assessment Test Questionnaire

SECONDARY OUTCOMES:
Changes in Anxiety and Depression Scale | Baseline and 12 weeks
  Evaluated by Hospital Anxiety and Depression Scale
Changes in Quality of Life Questionnaire | Baseline and 12 weeks
  Evaluated by self-reported Chronic Respiratory Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, Ph.D., Study Chair — University of Sao Paulo
Locations (1):
- Pulmonary and Rehabilitation Ambulatory of the Clinical Hospital of the University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Background] Donesky-Cuenco D, Nguyen HQ, Paul S, Carrieri-Kohlman V. Yoga therapy decreases dyspnea-related distress and improves functional performance in people with chronic obstructive pulmonary disease: a pilot study. J Altern Complement Med. 2009 Mar;15(3):225-34. doi: 10.1089/acm.2008.0389. PMID 19249998
- [Background] Brown RP, Gerbarg PL. Sudarshan Kriya yogic breathing in the treatment of stress, anxiety, and depression: part I-neurophysiologic model. J Altern Complement Med. 2005 Feb;11(1):189-201. doi: 10.1089/acm.2005.11.189. PMID 15750381
- [Background] Pomidori L, Campigotto F, Amatya TM, Bernardi L, Cogo A. Efficacy and tolerability of yoga breathing in patients with chronic obstructive pulmonary disease: a pilot study. J Cardiopulm Rehabil Prev. 2009 Mar-Apr;29(2):133-7. doi: 10.1097/HCR.0b013e31819a0227. PMID 19305239
- [Background] Santaella DF, Devesa CR, Rojo MR, Amato MB, Drager LF, Casali KR, Montano N, Lorenzi-Filho G. Yoga respiratory training improves respiratory function and cardiac sympathovagal balance in elderly subjects: a randomised controlled trial. BMJ Open. 2011 May 24;1(1):e000085. doi: 10.1136/bmjopen-2011-000085. PMID 22021757